CLINICAL TRIAL: NCT05114031
Title: FB101 Intervention in Asymptomatic Healthy Volunteers Who Have Undergone Vaginal Microbiome Screening - a Randomised, Double-blind, Placebo-controlled Study
Brief Title: FB101 Intervention in Women Screened to Have Vaginal Dysbiosis
Acronym: DYSCOVER-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freya Biosciences ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DYSCOVER-1
Record Dates: First submitted 2021-10-19; First posted 2021-11-09 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2021-10

CONDITIONS: Vaginal Flora Imbalance

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, parallel, 2-arm, placebo-controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, clinical investogators as well as outcome assessors (laboratories) will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FB101 (Experimental): Active intervention with microbial product FB101
  Interventions: Other: FB101
- Placebo (Placebo Comparator): Non-microbial placebo intervention
  Interventions: Other: Placebo

INTERVENTIONS:
Other: FB101 — Microbial intervention using product FB101
  Arms: FB101
Other: Placebo — Saline water
  Arms: Placebo

SUMMARY:
This study will explore and map the potential shifts in vaginal microbiomes as a consequence of a microbial intervention with product FB101 in healthy, asymptomatic volunteer women screened to have vaginal dysbiosis based on criteria defined by metagenomic sequencing of a vaginal swab sample.

DETAILED DESCRIPTION:
This study will explore and map the potential shifts in vaginal microbiomes as a consequence of a microbial intervention with product FB101 in healthy, asymptomatic volunteer women screened to have vaginal dysbiosis based on criteria defined by metagenomic sequencing of a vaginal swab sample. A dose of FB101 will be given on 3 different days and subjects will be followed for changes in their vaginal microbiomes until approximately 6 months after the first FD101 dose.

The study includes a screening visit where all criteria for participation are checked and a vaginal swab is obtained to check if pre-defined dysbiosis criteria are met based on metagenomic sequencing. If, and when, all criteria are confirmed, a baseline visit, visit 2, is scheduled to be performed around day 8 of the following menstrual cycle of each individual subject. Besides baseline assessments, the subject is randomised to active FB101 or placebo in a ratio of 3(active): 1(placebo) and the first dose is given. At visit 3 and 4 (performed on day 9 and 10 in the same menstrual cycle as Visit 2) the following 2 doses are given.

In total, 7 follow-up visits (visit 5-11) are scheduled to occur for a period of up to 6 months after the first dose. All follow-up visits will be scheduled to occur around day 8 in the subject's menstrual cycle with one menstrual cycle in between visits. At follow up visits, close safety monitoring will be performed as well as metagenomic sequencing assessment of the microbiota in a vaginal swab.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to give written informed consent.
* Age between ≥18 to ≤45.
* Is generally healthy, as determined by the investigator.
* Free of self-reported vaginal symptoms.
* Pre-menopausal women.
* Meets the following pre-defined criteria of vaginal dysbiosis: Combined Lactobacilli relative abundance below 10 % AND combined relative abundance of Gardnerella + Atopobium + Prevotella above 20 % based on metagenomic sequencing of vaginal sample.
* Has regular, predictable menstrual cycles of known length OR has been amenorrhoeic for at least 3 months due to use of a long-acting progestin or hormonal contraceptives.
* Is willing to be asked questions about personal medical, sexual, and behavioural history.
* Is willing to self-collect cervicovaginal secretions and vaginal swab samples at the clinic.
* Is willing to abstain from vaginal intercourse, unless using condoms, without the use of adjunctive spermicide or lubricant for at least one menstrual cycle length (28 days) after the intervention.
* Is willing to avoid taking baths, swimming, sitting in a hot tub, or wearing thong underwear for at least one menstrual cycle length (28 days) after the intervention.
* Is willing to abstain from using insertive vaginal feminine products (i.e., tampons, menstrual cups, sex toys), vaginal cleansing products, spermicides, lubricants, or other vaginal products not approved by the study investigators for at least 1 menstrual cycle length (28 days) after the intervention.

Exclusion Criteria:

* Participants who are post-menopausal, defined as more than 12 consecutive months of amenorrhea without another known cause than use of long-acting progestin or hormonal contraceptives.
* Participants who are pregnant, breastfeeding and/or have been pregnant within the last two months.
* Participants currently of childbearing potential, but not using an effective method of contraception, as outlined below:

  * Complete abstinence from intercourse two weeks prior to the intervention, throughout the clinical study, until the completion of follow-up procedures or for two weeks following discontinuation of the study participation in cases where participant discontinues the study prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
  * Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that participant.
  * Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), or contraceptive pill. The participant must be using this method for at least 1 week following the end of the study.
  * Use of any non-hormonal intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1 % per year. The participant must have the device inserted at least 3 months prior to the first Screening Visit, throughout the study, and 2 weeks following the end of the study.
* Women in same-sex relationships, or who are likely to engage in sexual relationships with other females throughout the study.
* Participants who have HIV/AIDS or other immunodeficiency.
* Participants who test positive at screening for HIV, chlamydia, gonorrhoea, Mycoplasma genitalium, and/or trichomonas vaginalis.
* Participants with a current vaginal candida infection, bacterial vaginosis or other condition requiring treatment that by the opinion of the investigator contraindicates participation in the current study.
* Participants may not be receiving treatment involving experimental drugs. If the participant has been in a recent experimental study, these must have been completed not less than 30 days prior to this study.
* Participants who have undergone some sort of procedure involving trauma to the cervix within the last 2 months prior to screening (i.e., IUD removal, cervical cryotherapy, or cervical laser treatment.
* Participants with any known condition requiring regular use of antibiotics, that would suggest the participant is likely to require antibiotic treatment during the study.
* Systemic and/or vaginally applied antibiotic use within the last month prior to screening.
* Participants with new (<3 months) use of long-acting hormonal treatments. Participant may be enrolled if stable (>3 months) or existing therapy as determined by the investigator.
* Participants with any social, medical, or psychiatric condition that in the opinion of the investigator would make it unlikely for the participant to comply with the study or would complicate interpretation of data from her participation.
* Participants with a history of drug or alcohol abuse that in the opinion of the investigator would make it unlikely for the participant to comply with the study or would complicate interpretation of data from her participation.
* Participants with a history of gynaecological cancers, gynaecological conditions, or surgical gynaecological medical history, which, in the opinion of the investigator, precludes participation.
* Participants with abnormal finding on screening exam, which, in the opinion of the investigator, precludes participation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in relative abundance of combined vaginal lactobacilli species | Comparing baseline (visit 2) to the following time points: 1 (visit 6), 2 (Visit 7), 3 (Visit 8), 4 (Visit 9), 5 (Visit 10) and 6 (Visit 11) months after Baseline
  The change in vaginal microbiome in active FB101 arm versus placebo arm measured as changes in relative abundance of combined vaginal lactobacilli species measured by metagenomic sequencing of vaginal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Fergus McCarthy, PHD, MD, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No